CLINICAL TRIAL: NCT07197788
Title: Endogenex Access Study
Brief Title: Continued Access to the Endogenex System for Participants in the ReCET Pivotal Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Endogenex, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1421
Record Dates: First submitted 2025-09-26; First posted 2025-09-29 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Type 2 Diabetes Mellitus; Type2diabetes; Diabetes Mellitus, Type 2; Type 2 Diabetes; Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Endogenex System Treatment (Experimental): Treatment arm will receive the Endogenex System procedure.
  Interventions: Device: Endogenex System

INTERVENTIONS:
Device: Endogenex System — The Endogenex System procedure utilizes a catheter to deliver non-thermal pulsed electric field to the first portion of the small intestine (duodenum) to induce cell regeneration. The catheter is introduced to the duodenum through the mouth using a guide wire and the therapy is applied to treat the duodenum.

SUMMARY:
This study is designed to collect real-world data on the safety and performance of the Endogenex System in the cohort of participants who were originally randomized to the sham control arm of the ReCET Study.

DETAILED DESCRIPTION:
This is a prospective, multicenter, open-label, treatment-only study designed to enroll individuals who participated in the ReCET Study, were randomized to the sham control arm, completed study follow-up, and are eligible, consented for participation in this study, and elect to receive treatment with the Endogenex System.

ELIGIBILITY:
Inclusion Criteria:

* Randomized to the sham control arm in the ReCET Study and completed their 12-month study visit.
* HbA1c of 7.0-10.5%, inclusive
* BMI <40 kg/m2, inclusive.
* Agree not to donate blood during participation in the study.
* Able to comply with study requirements and understand and sign the Informed Consent Form.
* Women of childbearing potential must be not pregnant and using an acceptable method of contraception throughout the study.
* Willing and able to comply with study visits and study tasks as required per protocol.

Exclusion Criteria:

* Diagnosed with type 1 diabetes.
* History of diabetic ketoacidosis or hyperosmolar nonketotic coma.
* Current use of insulin, or previous use of any types of insulin for >1 month at any time (except for treatment of gestational diabetes) in last 2 years.
* Hypoglycemic unawareness.
* History of ≥1 severe hypoglycemia episode in past 6 months
* Discontinuation of a GLP-1RA or a GLP-1/GIP dual-agonist within 6 months of the screening visit following at least one month of treatment.
* Known autoimmune disease, including but not limited to, celiac disease, or pre-existing symptoms of systemic lupus erythematosus, scleroderma or other autoimmune connective tissue disorder, or as evidenced by a positive anti-glutamic acid decarboxylase (GAD) test.
* Previous GI surgery that has changed GI anatomy or could limit treatment of the duodenum, such as Billroth 2, Roux-en-Y gastric bypass, gastric band or other similar procedures or conditions.
* Known history of a structural or functional disorder of the upper GI tract that may impede passage of the device through the upper GI tract or increase risk of tissue damage during an endoscopic procedure, including eosinophilic esophagitis, stricture/stenosis, varices, diverticula, or other disorder of the esophagus, stomach and duodenum.
* History of gastroparesis.
* Acute gastrointestinal illness in the last 7 days.
* Known history of irritable bowel syndrome, radiation enteritis or other inflammatory bowel disease, such as Crohn's disease and Celiac disease.
* History of chronic or acute pancreatitis.
* Active hepatitis or active liver disease, or alanine aminotransferase (ALT) level >3.0 times the upper limit of normal (ULN) for the reference range, as determined by the central laboratory at screening visit. Patients with NAFLD are eligible if their ALT level is ≤3.0 times the ULN.
* Current use of vitamin K antagonists such as warfarin, or current use of direct-action oral anticoagulants (DOCAs) that cannot be safely discontinued periprocedurally.
* Current use of P2Y12 inhibitors (clopidogrel, prasugrel, ticagrelor) that cannot be discontinued for 7 days before the procedure.
* Unable to discontinue non-steroidal anti-inflammatory drugs (NSAIDs) from treatment through 4 weeks following the procedure. Alternative use of acetaminophen and low dose aspirin is allowed.
* Use of systemic glucocorticoids (excluding topical or ophthalmic application or inhaled forms) for more than 10 consecutive days within 12 weeks prior to the screening visit.
* Use of medications known to affect GI motility (e.g. metoclopramide/ Reglan)
* Current use of weight loss medications such as Saxenda [liraglutide ], Xenical® [orlistat], Acutrim® [phenylpropanolamine], Sanorex® [mazindol], Adipex® [phentermine], BELVIQ® [lorcaserin], Qsymia® [phentermine/topiramate combination], Contrave® [naltrexone/bupropion], or other weight loss medications including over-the-counter [OTC] medications [for example, Allī®]) or have discontinued weight loss medications within 6 months.
* Participation in any structured weight loss program or endoscopic weight loss intervention within 6 months of the screen visit.
* Persistent anemia, defined as hemoglobin <10 g/dL.
* Known history of hemoglobinopathy, hemolytic anemia or sickle cell anemia, or any other traits of hemoglobin abnormalities known to interfere with the measurement of HbA1c.
* History of blood donation or transfusion within 3 months prior to the Screening Visit.
* Unstable or paroxysmal cardiac arrhythmia.
* Any of the following cardiovascular conditions within 6-months prior to screening visit: acute myocardial infarction, unstable angina, cerebrovascular accident (stroke), hospitalization due to congestive heart failure, or history of other significant cardiovascular disease (unless documented clearance by cardiologist and/or treating endoscopy team).
* History of valvular heart disease or chronic heart failure (NYHA III or IV).
* Estimated glomerular filtration rate (eGFR) ≤ 45 ml/min/1.73m2 calculated by CKD-EPI Creatinine Equation as determined by the central laboratory.
* Known immunocompromised status, including but not limited to individuals who have undergone organ transplantation, chemotherapy, or radiotherapy within the past 12 months, who have clinically significant leukopenia, who are positive for the human immunodeficiency virus (HIV) or whose immune status makes the participant a poor candidate for clinical trial participation in the opinion of the investigator.
* History of secondary hypothyroidism or inadequately controlled primary hypothyroidism (TSH value outside the normal range at screening).
* Presence of any implanted electronic devices that cannot be turned off during the procedure
* Presence of duodenal or biliary stents.
* Not a candidate for upper GI endoscopy or general anesthesia.
* Active illicit substance abuse or alcoholism (>2 drinks/day regularly).
* Active malignancy within the last 5 years (excluding non-melanoma skin cancers).
* Women who are breastfeeding.
* Participating in another ongoing clinical trial of an investigational drug or device.
* Binge eating disorder, or any other mental or physical condition which, in the opinion of the study investigator, makes the participant a poor candidate for clinical trial participation.
* Critically ill or has a life expectancy <5 years.
* Are investigator site personnel directly affiliated with this study and/or their immediate family member. Immediate family is defined as a spouse, parent, child, or sibling, whether biological or legally adopted.
* Uncontrolled hyperglycemia with a glucose level >270 mg/dl (>15 mmol/L) after an overnight fast or >360 mg/dl (>20 mmol/l) in a randomly performed measurement that is confirmed by a second measurement (not on the same day) at baseline or prior to the procedure.
* Any severe hypoglycemic event between baseline and the index procedure visits.
* Poorly controlled hypertension, as evidenced by a mean of 3 separate blood pressure measurements >180 mmHg (systolic) or >100 mmHg (diastolic)
* Women of child-bearing potential with a positive urine pregnancy test at baseline visit.
* LA Grade C or greater esophagitis on endoscopy.
* Abnormalities of the GI tract preventing endoscopic access to the duodenum.
* Anatomic abnormalities in the duodenum that would preclude the completion of the treatment procedure, including tortuous anatomy.
* Endoscopic observation of upper gastrointestinal abnormalities such as ulcers, duodenal polyps in the area to be treated, varices, strictures, congenital or intestinal telangiectasia.
* Any other anatomical or endoscopic abnormalities/characteristics that, in the opinion of the investigator, would preclude safe use of the investigational device or procedure.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2027-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events | 6 months post-procedure
  Incidence of device- and/or procedure-related serious adverse events

OTHER OUTCOMES:
Changes in glycemic control | 6 months post-procedure
  Change in HbA1c (%) from baseline to Month 6

IPD SHARING:
Plan to Share IPD: No